CLINICAL TRIAL: NCT06189690
Title: Effects of 5-Hz Repetitive Transcranial Magnetic Stimulation on Serum Brain Derived Neurotrophic Factor and Clinical Variables in Cocaine Use Disorder
Brief Title: Effect of HF rTMS on Serum BDNF in Cocaine Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Erik D. Morelos-Santana, Principal Investigator, Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMS-Coc-BDNF
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Cocaine Dependence
Keywords: Craving; BDNF; rTMS; DLPFC
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rTMS 5 Hz group (Experimental): Two-session/day 5-Hz rTMS will be administered by two week (weekdays) with a 30-minutes inter-session interval. A total of 20 sessions will be administered. Then two sessions per week along 12 weeks will be administered as maintenance phase. Parameters are considered as follow: 10 s. train, 10 s. inter-train interval, 2500 pulses per session at 100% of motor threshold (MT).
  Interventions: Device: rTMS
- Sham group (Sham Comparator): Two-session/day sham 5-Hz rTMS will be administered by two week (weekdays) with a 30-minutes inter-session interval. A total of 20 sessions will be administered. Then two sessions per week along 12 weeks will be administered as maintenance phase. Parameters are considered as follow: 10 s. train, 10 s. inter-train interval, 2500 pulses per session at 100% of motor threshold (MT).
  Interventions: Device: rTMS
- no rTMS control group (No Intervention): The patients on this group will receive any rTMS intervention. The purpose of this gruop is to compare all clinical, cognitive variables and BDNF levels under conditions of no cocaine/crack consumption, i.e., controlled environments, without rTMS.

INTERVENTIONS:
Device: rTMS — Repetitive TMS will be administered by a MagPro R30 stimulator and an active/placebo MCF-B70 A/P coil. All participants will use two surface electrodes to simulate rTMS skin sensations near to stimulation site. rTMS/sham conditions will be double-blinded by a USB stick. The USB contains the information about rTMS/sham condition and this is not available to the stimulator operator. Parameters of rTMS were previously described.
  Arms: Sham group; rTMS 5 Hz group

SUMMARY:
This study aims to explore the effect of 5-Hz rTMS over the left dorsolateral prefrontal cortex on the BDNF, craving and cognitive function. This study will be longitudinal, with a short-term double-blind placebo-controlled phase consisting of 20 rTMS sessions and a long-term phase, consisting of 2 weekly sessions for 12 weeks. Participants will be clinically assessed pre-treatment (T0), after 20-sessions phase (T1) and after 12-weeks phase (T2) by an interview about psychiatric symptoms. Also, blood will be obtained in the same T0, T1 and T2 to peripheral levels of BDNF determination. Cognitive state will be measured at the same time-points (T0, T1, T2) by paper-pencil and computerized neuropsychological assessment. Researchers will compare active rTMS versus placebo 5 Hz-rTMS on described variables. Additionally, a comparative group (without rTMS intervention) will be included to equivalently measure described variables during periods without cocaine consumption.

DETAILED DESCRIPTION:
Brain derived neurotrophic factor (BDNF) is a widely explored neurotrophin in preclinical models of cocaine addiction with relevant phase and region dependent dynamics along addictive cycle. In humans with cocaine use disorder (CUD), peripheral BDNF have revealed relationship with relevant treatment outcomes as relapse and time of abstinence. In CUD several interventional studies using high frequency repetititve transcranial magnetic stimulation (rTMS) have shown craving reduction, mood improvements and sustained modifications in functional conectivity measued by fMRI. Due to the relevance of BDNF in CUD, and neuroplasticity-related processes derived from rTMS interventions, this study aims to determine changes in peripheral BDNF, craving, cognition in CUD in reponse to rTMS. Aditionally, other outcomes will be considered as depression, anxiety and motivational changes.

Procedure: Psychiatric clinical and cognitive assessment, and blood collection will be performed at T0, T1 and T2 time-points. Short-term rTMS phase will consist of two weeks (weekdays) with 2 rTMS or rTMS-placebo sessions (detaills in arms section). Then, two sessions per week along 12 weeks as maintenance therapy will be considered. No rTMS group will attend the same time points and assessment in a controlled facility.

ELIGIBILITY:
Inclusion Criteria:

1. Current cocaine use disorder according to the Diagnostic and statistical manual of mental disorders (DSM 5).
2. Cocaine crack or powder use for at least 12 months with a frequency of 3 times or more per week, with abstinence periods shorter than 1 year for the last year.
3. Primary school completed.

Exclusion Criteria:

1. Personal or first degree family history of any neurological disorder including, but not limited to, organic brain syndrome, epilepsy, brain injuries, multiple sclerosis, conditions that increase intracranial pressure.
2. Personal history of brain surgery or traumatic brain injury.
3. Comorbilities that could represent a risk of neuroinfection or increased convulsive threshoid.
4. Other than alcohol, tobacco or marijuana substance use disorder.
5. If the patient does not meet the safety criteria for rTMS.
6. Current use of any medication that might provoque seizures or any anticonvulsant drugs.
7. Personal history of schizophrenia, mania/hypomania or OCD.
8. Personal history of myocardial infarction, angina, congestive heart failure, cerebrovascular events, transient ischemic attack or any other heart condition currently undergoing medical treatment.
9. Personal history of seizures or detection of paroxysmal EEG activity.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
BDNF | T0 before the intervention, T1: after rTMS 2 weeks, T2: after 12 weeks maintenance phase
  Serum BDNF levels will be measured by an ELISA kit following the manufacturer's instructions.
Cocaine craving | T0 before the intervention, T1: after rTMS 2 weeks, T2: after 12 weeks maintenance phase
  The Cocaine Craving Questionnaire (CCQ) in the general and now versions will be used to measure craving. Additionally, the visual analog scale (VAS) to cocaine/crack desire consumption will be used as craving measurement.

SECONDARY OUTCOMES:
Depression | T0 before the intervention, T1: after rTMS 2 weeks, T2: after 12 weeks maintenance phase
  The 17-item Hamilton Depression Rating Scale (HAM-D) will be used,
Anxiety | T0 before the intervention, T1: after rTMS2 weeks, T2: after 12 weeks maintenance phase
  The 14-item Hamilton Anxiety Rating Scale (HAM-A) will be used.

OTHER OUTCOMES:
Psychological problems | T0 before the intervention, T1: after rTMS2 weeks, T2: after 12 weeks maintenance phase
  The self-administered 90-item Symptoms Checklist-90 (SCL90) will be used.
Addiction severity | T0 before the intervention, T1: after rTMS2 weeks, T2: after 12 weeks maintenance phase
  The structured interview Addiction Severity Index Lite (ASI-Lite) wil be used to evaluate severity regarding the use of drugs and alcohol.
Previous cocaine-crack comsumption | T0 before the intervention, T1: after rTMS2 weeks, T2: after 12 weeks maintenance phase
  A retrospective calendar-based self report will be used to measure days of consumption previous to the study enrollment.
Motivation to change | T0 before the intervention, T1: after rTMS2 weeks, T2: after 12 weeks maintenance phase
  The 32-item self-administered form of University of Rhode Island Change Assessment (URICA) will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Psiquiatría Ramón de la Fuente M., Mexico City, Tlalpan, Mexico